CLINICAL TRIAL: NCT00422084
Title: A Phase III Comparative (Double-blind, Double-dummy) Randomised, Multi-centre Study to Assess the Efficacy of Pyronaridine Artesunate (180:60mg) Versus Coartem® (Artemether Lumefantrine) in Children & Adult Patients With Falciparum Malaria
Brief Title: Pyronaridine Artesunate (3:1) Versus Coartem® in P Falciparum Malaria Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medicines for Malaria Venture (Other)
Collaborators: Shin Poong Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SP-C-005-06
Record Dates: First submitted 2007-01-12; First posted 2007-01-15 (Estimated); Results first posted 2021-09-20 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Malaria
Keywords: malaria; antimalarial; artemisinin based combination therapy (ACT); P. falciparum; pyronaridine artesunate (Pyramax)
MeSH Terms: conditions — Malaria | interventions — pyronaridine tetraphosphate, artesunate drug combination; Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- PA group (Experimental): Pyronaridine artesunate (PA)
  Interventions: Drug: Pyronaridine artesunate
- AL group (Active Comparator): Arthemether lumefantrine (AL)
  Interventions: Drug: Coartem® (artemether lumefantrine)

INTERVENTIONS:
Drug: Pyronaridine artesunate — Oral PA (180:60mg tablets) once a day plus AL-placebo (twice a day) for 3 consecutive days (Day 0, 1, and 2)
  Other Names: Pyramax
  Arms: PA group
Drug: Coartem® (artemether lumefantrine) — AL (20:120mg tablets) twice a day plus PA-placebo (once a day) for 3 consecutive days (Day 0, 1, and 2)
  Other Names: Coartem
  Arms: AL group

SUMMARY:
The primary objective of this phase III study is to compare the efficacy and safety of the fixed combination of pyronaridine artesunate (Pyramax®, PA) with that of Coartem® (artemether lumefantrine, AL) in children and adults with uncomplicated P falciparum malaria in Africa and South East Asia.

DETAILED DESCRIPTION:
This is a multi-centre, comparative, randomised, (double-blind, double-dummy), parallel-group, non-inferiority study comparing the efficacy and safety of the fixed combination of PA with that of AL in the treatment of acute, uncomplicated P. falciparum malaria. The study population will include 1269 patients, comprising male and female children (≥20 kg body weight) and adults recruited from study sites in Africa and South East Asia.

Patients will be randomised to receive either oral PA (180:60mg tablets) once a day plus AL-placebo (twice a day) for 3 consecutive days (Days 0, 1, and 2) or AL twice a day plus PA-placebo (once a day) for 3 consecutive days (Days 0, 1, and 2) in a 2:1 ratio. The dose range of PA covered by this regimen is 7.2:2.4 mg/kg to 13.8:4.6 mg/kg, respectively, which has been shown to be effective and safe in Phase I and II studies. Posology will be based on body weight ranges for both the PA and AL regimens.

Patients will be confined to the study facility for ≥4 days (Days 0, 1, 2, and 3) and remain near the study site for ≥7 days, or once fever and parasite clearance has been confirmed for ≥24 hours - whichever occurs later.

The primary efficacy end point for the study is the proportion of patients with PCR-corrected adequate clinical and parasitological response (ACPR) on Day 28. Scheduled follow-up visits will continue until completion of the study at Day 42. In the case of adverse events reported and unresolved at Day 42, patients will be followed up for a further 30 days, or until resolution of the event.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients between the age of 3 and 60 years, inclusive.
* Body weight between 20 kg and 90 kg with no clinical evidence of severe malnutrition.
* Presence of acute uncomplicated P. falciparum mono-infection confirmed by:

  1. Fever, as defined by axillary/tympanic temperature ≥ 37.5°C or oral/rectal temperature ≥ 38°C, or documented history of fever in the previous 24 hours and,
  2. Positive microscopy of P. falciparum with parasite density between 1,000 and 100,000 asexual parasite count/μl of blood.
* Written informed consent, in accordance with local practice, provided by patient and/or parent/guardian/spouse.
* Ability to swallow oral medication.

Exclusion Criteria:

* Patients with signs and symptoms of severe/complicated malaria requiring parenteral treatment according to the World Health Organization Criteria 2000.
* Mixed Plasmodium infection.
* Severe vomiting or severe diarrhoea.
* Known history or evidence of clinically significant disorders.
* Presence of significant anaemia, as defined by Hb <8 g/dL.
* Presence of febrile conditions caused by diseases other than malaria.
* Known history of hypersensitivity, allergic or adverse reactions to pyronaridine, lumefantrine or artesunate or other artemisinins.
* Patients with known disturbances of electrolytes balance, e.g., hypokalaemia or hypomagnesaemia.
* Use of any other antimalarial agent within 2 weeks prior to start of the study as evidenced by a positive urine test.
* Female patients of child-bearing potential must be neither pregnant (as demonstrated by a negative pregnancy test) nor lactating, and must be willing to take measures to not become pregnant during the study period.
* Patients taking any drug which is metabolised by the cytochrome enzyme CYP2D6 (flecainide, metoprol, imipramine, amitriptyline, clomipramine).
* Received an investigational drug within the past 4 weeks.
* Known active Hepatitis A IgM (HAV-IgM), Hepatitis B surface antigen. (HBsAg) or Hepatitis C antibody (HCV Ab).
* Known seropositive HIV antibody.
* Liver function tests [ASAT/ALAT levels] >2.5 times the upper limit of normal range.
* Known significant renal impairment as indicated by serum creatinine >1.4 mg/dL.

Ages: 3 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1272 (Actual)
Dates: Start 2007-01; Primary Completion 2008-04 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claude Oeuvray, PhD, Study Director — Medicines for Malaria Venture
Locations (10):
- Ecole de Santé Publique, Faculté de Médecine, Université de Kinshasa, Kinshasa, Democratic Republic of the Congo
- Komfo Anoykye Teaching Hospital, Kumasi, Ghana
- Indonesia (2):
  - RSUD TC Hillers, Maumere, Nusa Tenggara Timur
  - Jayapura General Hospital (RSUD) DOK II, Jayapura, Special Region of Papua
- Siaya District Hospital, Medical Superintendent's office, Siaya, Kenya
- Malaria Research and Training Center, Faculté de Médecine, de Pharmacie et d'Ondonto-stomatologie, Bamako, Mali
- Instituto Nacional de Saude, Ministero de Saude, Maputo, Mozambique
- Puerto Princesa General Hospital, Puerto Princesa City, Philippines
- Service de Parasitologie, Faculté de Médecine, Université Cheikh Anta Diop, Dakar, Dakar Fann, Senegal
- Farafenni Field Station, c/o: MRC Laboratories, Fajara, The Gambia

REFERENCES:
- [Result] Tshefu AK, Gaye O, Kayentao K, Thompson R, Bhatt KM, Sesay SS, Bustos DG, Tjitra E, Bedu-Addo G, Borghini-Fuhrer I, Duparc S, Shin CS, Fleckenstein L; Pyronaridine-artesunate Study Team. Efficacy and safety of a fixed-dose oral combination of pyronaridine-artesunate compared with artemether-lumefantrine in children and adults with uncomplicated Plasmodium falciparum malaria: a randomised non-inferiority trial. Lancet. 2010 Apr 24;375(9724):1457-67. doi: 10.1016/S0140-6736(10)60322-4. PMID 20417857
- [Derived] Pryce J, Taylor M, Fox T, Hine P. Pyronaridine-artesunate for treating uncomplicated Plasmodium falciparum malaria. Cochrane Database Syst Rev. 2022 Jun 21;6(6):CD006404. doi: 10.1002/14651858.CD006404.pub4. PMID 35726133
- [Derived] Ayyoub A, Methaneethorn J, Ramharter M, Djimde AA, Tekete M, Duparc S, Borghini-Fuhrer I, Shin JS, Fleckenstein L. Population Pharmacokinetics of Pyronaridine in Pediatric Malaria Patients. Antimicrob Agents Chemother. 2015 Dec 14;60(3):1450-8. doi: 10.1128/AAC.02004-15. PMID 26666916
- [Derived] Duparc S, Borghini-Fuhrer I, Craft CJ, Arbe-Barnes S, Miller RM, Shin CS, Fleckenstein L. Safety and efficacy of pyronaridine-artesunate in uncomplicated acute malaria: an integrated analysis of individual patient data from six randomized clinical trials. Malar J. 2013 Feb 21;12:70. doi: 10.1186/1475-2875-12-70. PMID 23433102

RESULTS

PARTICIPANT FLOW:
Groups:
- AL Group: Arthemether lumefantrine (AL)
  Coartem® (artemether lumefantrine): AL twice a day plus PA-placebo (once a day) for 3 consecutive days (Day 0, 1, and 2)
Period: Overall Study
Arm/Group | PA Group | AL Group
Started | 849 | 423
Completed | 751 | 347
Not Completed | 98 | 76
Not completed — Adverse Event | 21 | 7
Not completed — Withdrawal by Subject | 12 | 9
Not completed — Lost to Follow-up | 14 | 9
Not completed — Protocol Violation | 4 | 1
Not completed — Lack of Efficacy | 40 | 42
Not completed — P. vivax infection | 3 | 6
Not completed — Cyesis | 1 | 0
Not completed — Withdrawn from study accidentally | 1 | 0
Not completed — Non-compliance | 1 | 0
Not completed — Re-location | 0 | 1
Not completed — Not defined | 1 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population, defined as all randomized subjects who received any amount of study medication. Subjects were analyzed as randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | PA Group | AL Group | Total
Number analyzed (Participants) | 849 | 423 | 1272
Age, Continuous [Mean (Standard Deviation); unit: years] | 17.2 (11.12) | 18.0 (11.41) | 17.5 (11.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 359 | 192 | 551
  Male | 490 | 231 | 721
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 722 | 358 | 1080
  Asian/Oriental | 127 | 65 | 192
Region of Enrollment [Number; unit: participants]
  Mozambique | 89 | 44 | 133
  Gambia | 72 | 34 | 106
  Mali | 132 | 66 | 198
  Senegal | 138 | 68 | 206
  Philippines | 67 | 36 | 103
  Congo, The Democratic Republic of the | 199 | 99 | 298
  Ghana | 4 | 3 | 7
  Kenya | 88 | 44 | 132
  Indonesia | 60 | 29 | 89

OUTCOME MEASURES:

1. Primary Outcome: PCR-Corrected Adequate Clinical and Parasitological Response (ACPR) Rate on Day 28
Description: Percentage of subjects with PCR-corrected adequate clinical and parasitological response (ACPR) on Day 28, defined as absence of parasitaemia on Day 28 without the subject's meeting any of the criteria of early treatment failure, late clinical failure, or late parasitological failure.
Time Frame: Day 28
Population: Efficacy evaluable population subjects completed a full course of study medication; has a known primary efficacy endpoint at D28; did not miss a dose due to vomiting (except at D0); did not use a concomitant medication (except acetaminophen); did not have a concomitant disease which may have interfered with the classification of the treatment outcome; and did not have major protocol deviations.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | PA Group | AL Group
Number analyzed (Participants) | 784 | 386
percentage of subjects | 99.5 [98.7 to 99.9] | 99.2 [97.7 to 99.8]
Statistical Analysis 1: Comparison: PA Group vs AL Group; Null hypothesis: The PCR-corrected ACPR response rate at Day 28 for the PA group is inferior to the PCR-corrected ACPR response rate at Day 28 for the comparator group (AL) by more than 5%. Was tested versus the alternative: Alternative hypothesis: The PCR-corrected ACPR response rate at Day 28 for the PA group is not inferior to the PCR-corrected ACPR response rate at Day 28 for the comparator group (AL) by more than -5%; Test type: Non-Inferiority or Equivalence — The primary efficacy analysis tested the non-inferiority of the PA group compared to the comparator group with regard to the PCR-corrected ACPR response rate at Day 28 using the 2-sided 95% confidence interval (CI) (Newcombe-Wilson score method without continuity correction) and a 5% non-inferiority margin. Non-inferiority was demonstrated if the lower limit of the CI for the difference >-5%; p = 0.578, Chi-squared — If non-inferiority of PA is demonstrated, the p-value associated with a superiority test was calculated based on a 2-sided Chi-square test. If the calculated p-value is <5%, then the superiority of PA compared to AL is statistically demonstrated; ACPR percent difference = 0.3, 95% CI 2-sided [-0.7 to 1.8]

2. Secondary Outcome: PCR-corrected Adequate Clinical and Parasitological Response (ACPR) on Day 14
Description: Percentage of subjects with PCR-corrected adequate clinical and parasitological response (ACPR) on Day 14, defined as absence of parasitaemia on Day 14 without the subject's meeting any of the criteria of early treatment failure, late clinical failure, or late parasitological failure.
Time Frame: Day 14
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | PA Group | AL Group
Number analyzed (Participants) | 784 | 386
percentage of subjects | 99.9 [99.3 to 100.0] | 100 [99.0 to 100.0]

3. Secondary Outcome: Crude ACPR (Non-PCR Corrected ACPR) on Day 14 and Day 28
Description: Percentage of subjects with adequate clinical and parasitological response (ACPR) on Day 28, without correction by PCR, defined as absence of parasitaemia on Day 28 without the subject's meeting any of the criteria of early treatment failure, late clinical failure, or late parasitological failure.
Time Frame: Day 14 and 28
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | PA Group | AL Group
Number analyzed (Participants) | 784 | 386
percentage of subjects
  Cure rate (%) at Day 14 | 100 [99.5 to 100.0] | 100 [99.0 to 100.0]
  Cure rate (%) at Day 28 | 98.9 [97.8 to 99.5] | 97.2 [95.0 to 98.6]

4. Secondary Outcome: Parasite Clearance Time
Description: Parasite clearance time is defined as the time from first dosing to the time of first blood draw with parasite clearance. Parasite clearance is defined as zero presence of asexual parasites for 2 consecutive negative readings taken between 7 and 25 hours apart.
Time Frame: Days 0, 3, 7, 14, 21, 28, 35, and 42 (or on any other day if the subject spontaneously returned)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | PA Group | AL Group
Number analyzed (Participants) | 784 | 386
hours | 23.9 [23.9 to 23.9] | 24.0 [23.9 to 24.1]

5. Secondary Outcome: Fever Clearance Time
Description: Fever clearance time is defined as the time from first dosing to first normal reading of temperature for 2 consecutive normal temperature readings taken between 7 and 25 hours apart
Time Frame: Day 0 and every 8 hours over ≥72 hours following first study drug administration or temperature normalization for ≥2 readings between 7 and 25 hours apart, then at each visit and as clinically indicated
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | PA Group | AL Group
Number analyzed (Participants) | 584 | 299
hours | 7.9 [7.9 to 8.0] | 8.0 [7.9 to 15.5]

6. Secondary Outcome: Percentage of Patients With Fever Clearance at Day 1, 2 and 3
Description: as for outcome 5
Time Frame: Days 1, 2, 3
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | PA Group | AL Group
Number analyzed (Participants) | 584 | 299
percentage of subjects
  Clearance rate (%) at Day 1 (24h after first dose) | 88.7 [86.0 to 91.1] | 87.0 [82.9 to 90.5]
  Clearance rate (%) at Day 2 (48h after first dose) | 99.0 [97.9 to 99.6] | 98.7 [96.8 to 99.6]
  Clearance rate (%) at Day 3 (72h after first dose) | 99.5 [98.6 to 99.9] | 99.3 [97.8 to 99.9]

7. Secondary Outcome: Proportion of Patients With Parasite Clearance at Day 1, 2 and 3
Description: Parasite clearance time is defined as the time from first dosing to the time of first blood draw with parasite clearance. Parasite clearance was defined as zero presence of asexual parasites for 2 consecutive negative readings taken between 7 and 25 hours apart.
Time Frame: Days 1, 2, 3
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | PA Group | AL Group
Number analyzed (Participants) | 784 | 386
percentage of subjects
  Clearance rate (%) at Day 1 (24h after first dose) | 68.1 [64.8 to 71.3] | 52.8 [48.0 to 57.9]
  Clearance rate (%) at Day 2 (48h after first dose) | 98.1 [96.9 to 98.9] | 97.2 [95.1 to 98.5]
  Clearance rate (%) at Day 3 (72h after first dose) | 99.5 [98.8 to 99.8] | 99.7 [98.6 to 100]

8. Secondary Outcome: Adverse Events and Clinically Significant Laboratory Results
Description: Incidence of adverse events and of clinically significant laboratory results, ECG, vital signs or physical examination abnormalities.
Time Frame: Day 0 to 42. Subjects experiencing AEs at Day 42 were followed for up to 30 days after the end of study or resolution of the event, whichever was earlier
Population: The safety population consists of all randomized subjects who received any amount of study medication; subjects were analyzed as treated.
Measure: Count of Participants; unit: Participants
Arm/Group | PA Group | AL Group
Number analyzed (Participants) | 849 | 423
Participants
  Nr subj. with ≥1 AE | 509 | 241
  Nr subj. with ≥1 treatment-related AE | 275 | 123
  Nr subj. with ≥1 SAE | 3 | 2
  Nr pat with ≥1 treatment-related SAE | 0 | 0
  Nr subj. with ≥1 severe or life-threatening AE | 10 | 5
  Nr subj. with ≥1 AE leading to death | 0 | 0
  Nr subj. ≥1 AE leading to drug discontinuation | 16 | 5
  Nr subj. with ≥1 AE leading to study withdrawal | 19 | 6

ADVERSE EVENTS:
Time Frame: Day 0 to 42. Subjects experiencing AEs at Day 42 were followed for up to 30 days after the end of study or resolution of the event, whichever was earlier
Description: An AE was defined as any unfavorable and unintended sign, symptom, syndrome, or illness that developed or worsened during the period of observation in the clinical study.
Arm/Group | PA Group | AL Group
All-Cause Mortality (participants affected / at risk) | 0/849 | 0/423
Serious Adverse Events (participants affected / at risk) | 3/849 | 2/423
Other Adverse Events (participants affected / at risk) | 506/849 | 239/423
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PA Group (N=849) | AL Group (N=423)
Parotitis (Infections and infestations) | 1 (1) | 0 (0)
Typhoid fever (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Cerebral malaria (Infections and infestations) | 0 (0) | 1 (1)
Immunosuppression (Immune system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PA Group (N=849) | AL Group (N=423)
Anaemia (Blood and lymphatic system disorders) | 17 (17) | 4 (4)
Eosinophilia (Blood and lymphatic system disorders) | 60 (60) | 26 (26)
Lymphocytosis (Blood and lymphatic system disorders) | 21 (23) | 16 (17)
Neutropenia (Blood and lymphatic system disorders) | 41 (45) | 27 (27)
Bradycardia (Cardiac disorders) | 5 (5) | 5 (5)
Vertigo (Ear and labyrinth disorders) | 14 (15) | 6 (6)
Abdominal pain (Gastrointestinal disorders) | 50 (50) | 23 (23)
Abdominal pain upper (Gastrointestinal disorders) | 13 (13) | 9 (10)
Diarrhoea (Gastrointestinal disorders) | 17 (17) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 9 (9) | 4 (4)
Nausea (Gastrointestinal disorders) | 14 (14) | 9 (9)
Toothache (Gastrointestinal disorders) | 9 (9) | 2 (2)
Vomiting (Gastrointestinal disorders) | 42 (43) | 15 (15)
Influenza like illness (General disorders) | 30 (30) | 13 (15)
Pyrexia (General disorders) | 20 (20) | 10 (10)
Helminthic infection (Infections and infestations) | 13 (13) | 6 (6)
Influenza (Infections and infestations) | 7 (7) | 8 (8)
Nasopharyngitis (Infections and infestations) | 13 (15) | 5 (5)
Oral herpes (Infections and infestations) | 16 (16) | 8 (8)
Respiratory tract infection (Infections and infestations) | 10 (12) | 2 (2)
Rhinitis (Infections and infestations) | 10 (10) | 9 (9)
Upper respiratoty tract infection (Infections and infestations) | 32 (36) | 12 (12)
Urinary tract infection (Infections and infestations) | 20 (21) | 9 (9)
Alanine aminotransferase increased (Investigations) | 9 (9) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 21 (23) | 6 (6)
Platelet count increased (Investigations) | 16 (19) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 8 (8) | 8 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 10 (10) | 2 (2)
Headache (Nervous system disorders) | 71 (76) | 41 (42)
Haematuria (Renal and urinary disorders) | 11 (11) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 49 (52) | 27 (27)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No